CLINICAL TRIAL: NCT07017777
Title: A Phase III, Observer-blind, Randomized Controlled Trial to Evaluate the Immunogenicity and Safety of 13-valent Pneumococcal Conjugate Vaccine (PCV13i) in Healthy Infants Aged 2 Months (Minimum 6 Weeks)
Brief Title: A Study to Evaluate the Immunogenicity and Safety of 13-valent Pneumococcal Conjugate Vaccine (PCV13i) in Healthy Infants Aged 2 Months (Minimum 6 Weeks)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CanSino Biologics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTP-PCV-002
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-05

CONDITIONS: Pneumococcal Infections; Streptococcal Infections; Bacterial Infections
Keywords: PCV13i; 13 valent Pneumococcal conjugate vaccine; Pneumococcal infections; 2 months of age; Safety; Immunogenicity
MeSH Terms: conditions — Pneumococcal Infections; Streptococcal Infections; Bacterial Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 13-valent Pneumococcal Polysaccharide Conjugate Vaccine (CRM197/TT) (PCV13i) (Experimental): Intramuscular Injection, 0.5ml
  Interventions: Biological: PCV13i
- Pneumococcal 13-valent Conjugate Vaccine (Prevnar 13) (Active Comparator): Intramuscular Injection, 0.5ml
  Interventions: Biological: Prevnar 13

INTERVENTIONS:
Biological: PCV13i — 3 doses: 2 months (Dose 1) months (Dose 2), 12-15 months (Booster dose)
  Arms: 13-valent Pneumococcal Polysaccharide Conjugate Vaccine (CRM197/TT) (PCV13i)
Biological: Prevnar 13 — 3 doses: 2 months (Dose 1) months (Dose 2), 12-15 months (Booster dose)
  Arms: Pneumococcal 13-valent Conjugate Vaccine (Prevnar 13)

SUMMARY:
This is a Phase 3 randomized, observation-blinded, active-controlled, parallel-group clinical trial designed to evaluate the immunogenicity, safety, and functional antibody response of the experimental vaccine versus the control vaccine in healthy Thailand infants vaccinated at a 2+1 schedule (2 months, 4 months and 12-15 months). The trial will enroll approximately 600 healthy infants aged 2 months (at least 6 weeks) who will be randomly assigned in a 1:1 ratio to receive either the experimental or control vaccine, with 100 in each group (200 in total) randomized to subgroups and subject to additional immunogenicity assessments. All participants will be evaluated for solicited adverse events for 7 days and unsolicited adverse events for 30 days post each vaccination. Immunogenicity evaluation will be performed in all participants at baseline and post the booster dose, while the sub-cohort participants will be evaluated for post primary series immunogenicity additionally.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants with stable clinical conditions aged 2 months (42-90 days) at the time of screening, based on medical history and clinical assessment by the investigator. Infants will be eligible starting from the day they turn 6 weeks of age.
* Infant's parent or legal guardian must be able and willing to provide informed consent for the infant's participation in the study.
* Participants and their parent or legal guardian must demonstrate the ability to comply with all trial procedures and be available for the entire follow-up duration.
* The infant's parent or legal guardian must have an easily identifiable and stable place of residence within the study area, be available for the duration of trial participation, and have access to a reliable means of telephone contact for communication with the study team.

Exclusion Criteria for the first dose:

* Infants born at <35 weeks of gestation.
* Infants who have previously received any pneumococcal vaccine.
* Infants currently participating in or who have recently participated in another interventional clinical trial.
* Infants with an axillary temperature of ≥37.8°C at the time of enrollment (the participant must be deferred until recovery. The visit may be rescheduled when this criterion is met.)
* Infants with any congenital abnormalities, chronic medical conditions, or genetic disorders, severe malnutrition, inherited disease and others, that in the investigator's judgment, may interfere with the study outcomes.
* History of anaphylactic shock
* History of allergic disease or history of a serious reaction to any prior vaccination or known hypersensitivity to any component of the experimental and control vaccine
* History of epilepsy and convulsions.
* Have received immunosuppressive treatment, cytotoxic treatment, systemic steroid treatment for more than 2 weeks, etc. (excluding local treatment, surface treatment of acute non-concurrent dermatitis, or spray treatment of allergic rhinitis).
* Received or planned to receive blood/plasma products or immunoglobulins throughout the study period or prior to study vaccination.
* History of coagulation disorders or blood conditions that could cause anemia or excess bleeding as judged by the investigator.
* Infants with known or suspected immunodeficiency, as determined by medical history and/or physical examination.
* Administration of other vaccines within 7 days prior to enrollment.
* Any history or current evidence of a condition or therapy that could confound study results, interfere with participation, or is not in the best interest of the participant, as judged by the investigator.
* The participant is a direct descendant (child or grandchild) of any person employed by the Sponsor, the contract research organization (CRO), the investigator, or study site personnel.
* Any other condition or situation that, in the investigator's judgment, might interfere with the study or pose additional risks to the participant.

Individual termination criteria for subsequent doses:

* Severe allergic reaction after the previous vaccination.
* Serious adverse events caused by the previous vaccination that is not suitable for subsequent vaccination(s) as judged by the investigator.
* Newly identified symptoms or newly occurred cases after the first vaccination that do not meet the inclusion criteria for the first dose, or that meet the exclusion criteria for the first dose. The decision to discontinue participation is determined by the investigator.
* Other reasons for exclusion considered by the investigator.

Ages: 6 Weeks to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 600 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving serotype-specific IgG antibody concentrations ≥ 0.35 µg/mL | 30 days after the booster dose
Incidence of solicited local and systemic adverse events (AEs) | Within 7 days after each dose of vaccination

SECONDARY OUTCOMES:
Incidence of unsolicited adverse events | Within 30 days after each dose of vaccination
The number of serious adverse events (SAEs) | Through study completion, an average of 16-19 months
The geometric mean concentration (GMC) of Serotype-specific IgG in all participants | Before vaccination and 30 days after the booster dose
Proportion of participants achieving serotype-specific IgG antibody concentrations ≥ 0.35 µg/mL in Sub-cohort A participants | 30 days after the primary series
Proportion of participants achieving serotype-specific IgG antibody concentrations ≥ 0.35 µg/mL in Sub-cohort B participants | Before the booster dose
The geometric mean concentration (GMC) of Serotype-specific IgG in Sub-cohort A participants | 30 days after the primary series
The geometric mean concentration (GMC) of Serotype-specific IgG in Sub-cohort B participants | Before the booster dose

CONTACTS AND LOCATIONS:
Overall Officials: Supattra Rungmaitree, Doctor of Medicine, Principal Investigator — Department of Pediatrics, Faculty of Medicine Siriraj Hospital, Mahidol University